CLINICAL TRIAL: NCT05034237
Title: The Effect of Long-pulsed 1064 nm nd: Yag Laser-assisted Hair Removal on Some Skin Flora and Pathogens: an in Vivo Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, marwa eldeeb, lecturer of dermatology, Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0106624
Record Dates: First submitted 2021-07-23; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Changes in Bacterial Count in Axilla After Laser Hair Removal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ND;YAG 1064 NM LASER (Experimental): monthly sessions of laser hair removal
  Interventions: Device: ND;YAG 1064NM LASER

INTERVENTIONS:
Device: ND;YAG 1064NM LASER — laser hair removal sessions

SUMMARY:
1. To evaluate the effect of ND-YAG laser hair removal on some skin flora and pathogens: an in vivo study.
2. To determine the immediate and long term effect of ND-YAG laser on total viable bacterial count, some skin flora and pathogens of laser-assisted hair removal in axilla.
3. To assess the relation between this effect and bromohidrosis.

DETAILED DESCRIPTION:
This Quasi-experimental interrupted time series study will be conducted on 30 female participants who will be recruited from the Dermatology Outpatient Clinic of the Alexandria Main University Hospital.

Four sessions of laser assisted hair removal at 4 weeks intervals (S1, S2, S3 and S4) using long pulsed ND: YAG (Cynosure Elite+™, Westford, USA). The following parameters will be used according to the nature of hair (1064 nm, 15-18 mm spot size, fluence of 24-35 J/cm2, pulse duration 30-40 ms).

4. Swabs will be collected immediately and after each session

ELIGIBILITY:
Inclusion Criteria:

No previous laser hair removal sessions involving axilla. Fitzpatrick skin type III-VI.

Exclusion Criteria:

1. Skin diseases such as atopic dermatitis, psoriasis, fungal or herpetic infections.
2. Systemic diseases such as diabetes or endocrinal dysfunction.
3. Patients receiving immunosuppressive therapy.
4. Pregnant or lactating females.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-14 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
to compare changes in bacterial count and composition of axillary flora after laser hair removal | 4 month
  counting bacterial colonies (aerobic,anaerobic,lipophyllic and staphylococcal) using colony counter

SECONDARY OUTCOMES:
To determine the immediate and long term effect of ND-YAG laser on total viable bacterial count, some skin flora and pathogens of laser-assisted hair removal in axilla | 4 month
  counting bacterial colonies immediately before and immediately after each laser session
To assess the relation between this effect and bromohidrosis. | 4 month
  using a questionnaire that is categorized into better , worse or unchanged sweat odour.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No